CLINICAL TRIAL: NCT05357846
Title: Phase III Multicenter Randomized Controlled Trial of PD-1 Inhibitor Combined With Preoperative Concurrent Chemoradiotherapy and Surgery for Locally Advanced Esophageal Squamous Cell Carcinoma (NEOCRTEC2101)
Brief Title: PD-1 Inhibitor Combined With Neoadjuvant Chemoradiotherapy Plus Surgery for Locally Advanced ESCC (NEOCRTEC2101)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Yang Hong, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOCRTEC2101
Record Dates: First submitted 2022-03-22; First posted 2022-05-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Esophageal Carcinoma; Esophageal Cancer; Oesophageal Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — sintilimab; Paclitaxel; Cisplatin; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NCRT+IO group (Experimental): • NCRT+IO group consists of the PD-1 inhibitor combined with concurrent chemoradiotherapy prior to surgery. The patient will receive 4 weeks of radiation therapy. The radiation will generally commence on the 1st day of treatment and will run for 4 weeks.PD-1 inhibitor is given by intravenous infusion on days 1 and 22. Chemotherapy is given by intravenous infusion on days 1, 8, 15, and 22.
  Interventions:
  * Radiation: (40 or 45 Gy/20 fractions)
  * Drug: Sintilimab
  * Drug: Paclitaxel
  * Drug: Cisplatin
  Interventions: Drug: Sintilimab; Radiation: Preoperative radiotherapy; Drug: Paclitaxel; Drug: Cisplatin; Procedure: esophagectomy
- NCRT group (Active Comparator): • NCRT group consists of the concurrent chemoradiotherapy prior to surgery. The patient will receive 4 weeks of radiation therapy. The radiation will generally commence on the 1st day of treatment and will run for 4 weeks. Chemotherapy is given by intravenous infusion on days 1, 8, 15, and 22.
  Interventions:
  * Radiation: (40 or 45 Gy/20 fractions)
  * Drug: Paclitaxel
  * Drug: Cisplatin
  Interventions: Radiation: Preoperative radiotherapy; Drug: Paclitaxel; Drug: Cisplatin; Procedure: esophagectomy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg, IV (in the vein) on day 1 and day 22
  Arms: NCRT+IO group
Radiation: Preoperative radiotherapy — External radiation with a total dose of 40.0 or 45.0 Gy is given in 20 fractions,5 fractions a week.
Drug: Paclitaxel — 50mg/m2, IV (in the vein) on day 1,day 8,day 15 and day 22
  Other Names: Taxol
Drug: Cisplatin — 25mg/m2,IV DRIP on day 1,day 8,day 15 and day 22
  Other Names: DDP
Procedure: esophagectomy — McKeown esophagectomy, Ivor Lewis esophagectomy or minimally invasive esophagectomy will be performed 6-8 weeks after chemoradiotherapy. Two-field lymphadenectomy with total mediastinal lymph node dissection is performed during surgery.

SUMMARY:
The primary objective is to compare PD-1 inhibitor combined with preoperative chemoradiotherapy followed by surgery versus neo-adjuvant chemoradiotherapy followed by surgery, in terms of the overall survival time (OS) in patients with Stage T1-4aN1-3M0 or T3-4aN0M0 squamous cell esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage T1-4aN1-3M0 or T3-4aN0M0,which is potentially resectable.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival.
4. Age ranges from 18 to 70 years.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. WHO PS score 0-1
7. Signed informed consent document on file.

Exclusion Criteria:

1. Patients have received any prior anticancer therapy.
2. Patients are diagnosed or suspected to be allergic to sintilimab,toxal or cisplatin.
3. Patients with concomitant hemorrhagic disease.
4. Patients who cannot tolerate surgery.
5. Pregnant or breast feeding.
6. Patients without informed consent because of psychological, family, social or any other factors.
7. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more.
8. Patients with malignant tumors other than esophageal cancer,except for non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer.
9. Patients with history of diabetes over 10 years and unsatisfactory glycemic control.
10. Patients with severe heart,lung,liver,renal dysfunction, hematopoietic system diseases, immune system diseases, cachexia or other diseases that lead to intolerance of chemoradiotherapy or surgery.
11. Patients with history of autoimmune diseases, immunodeficiency, or organ and allogeneic bone marrow transplantation.
12. Patients with history of interstitial lung disease or noninfectious pneumonia.
13. Patients with active pulmonary tuberculosis infection, or a history of active pulmonary tuberculosis infection within one year before enrollment, or a history of active pulmonary tuberculosis infection more than one year ago without regular treatment.
14. Patients with active hepatitis B ( HBV DNA ≥ 2000 IU / mL or 104 copies / mL ) or hepatitis C ( HCV antibody positive ).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At end of enrollment- up to 5 years in follow up
  Overall survival will be calculated from the date of randomization and an event registered on the date of death from any cause. Patients lost to follow up, or those with no death recorded on the day the database is frozen, will be censored on the date of last follow up.

SECONDARY OUTCOMES:
Progression free survival | At end of enrollment- up to 5 years in follow up
  Progression free survival is defined as the time from randomization until objective tumor progression or death.
Pathologic complete response rate | Two weeks after surgery
  No malignant tumor cells were detected in the removed specimens including primary tumor and lymph nodes
R0 resection rate | Two weeks after surgery
  The percentage of patients who undergo complete resection
Incidence of perioperative complications | Ninety days after surgery
  Incidence of complications
Perioperative mortality | Ninety after surgery
  Incidence of death postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: HONG YANG, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No